CLINICAL TRIAL: NCT07303582
Title: Individualised Cryoneurolysis to Treat Pain in the Context of Spasticity in the Upper and Lower Extremities (ICE): a Pilot Randomised Controlled Trial
Brief Title: Individualised Cryoneurolysis to Treat Pain in the Context of Spasticity in the Upper and Lower Extremities
Acronym: ICE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: University of Oxford (Other); Bournemouth University (Other)
Responsible Party: Principal Investigator, Anton Pick, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PID 18403
Record Dates: First submitted 2025-09-10; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Centreal Neurological Condition; Acquired Brain Injury (Including Stroke); Multiple Sclerosis; Spinal Cord Injury
Keywords: Cryoneurolysis; Spasticity; Pain; Acquired Brain Injury; Stroke; Multiple Sclerosis; Spinal Cord Injury; Central Neurological Condition; Botulinum Toxin (botox); Iovera; Chemodenervation; BoNT-A; Cryoneurotomy; Cryoneurectomy; Cryoanalgesia
MeSH Terms: conditions — Brain Injuries; Multiple Sclerosis; Spinal Cord Injuries; Muscle Spasticity; Pain; Stroke | interventions — Botulinum Toxins; Botulinum Toxins, Type A; incobotulinumtoxinA; Nerve Block

STUDY DESIGN:
Intervention Model Description: Participants randomised to control will be given the opportunity (but are not required) to crossover to the intervention arm at 12-weeks post-treatment. The intervention arm will not crossover to control arm.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoneurolysis (+ usual care) (Experimental)
  Interventions: Procedure: Cryoneurolysis
- Botulinum Toxin (+ usual care) (Active Comparator)

INTERVENTIONS:
Procedure: Cryoneurolysis — Nerves that require treatment, and the number of treatments required for each nerve will be identified by routine clinical judgement. Nerve targets are identified using an ultrasound machine. The handheld Iovera cryoneurolysis device will be used for treatment.
  Participants will receive up to 4 treatments of cryoneurolysis for each nerve or nerve branch that requires treatment. It is anticipated that participants will have between 1 and 5 nerves or nerve branches per limb treated. Each Cryoneurolysis treatment takes 110 seconds. Total treatment time will be determined by number of nerves targeted and number of cryoneurolysis treatments per nerve. The shortest duration, with setup, is likely to be 60 minutes and the longest 120 minutes.
  Other Names: Iovera; Cryoneurotomy; Cryoneurectomy; Cryoanalgesia
  Arms: Cryoneurolysis (+ usual care)
Procedure: Botulinum toxin — Muscles that require treatment with Botulinum Toxin will be identified by routine clinical assessment. Muscle targets will be identified using an ultrasound machine.
  It is anticipated that participants will have between 2 and 8 muscles identified for target. The participant will receive up to 200 units of Xeomin (Botulinum Toxin) per muscle that requires treatment. Treatment session of Botulinum Toxin will take 60 to 90 minutes.
  Other Names: Botox; Xeomin; Chemodenervation; BoNT-A

SUMMARY:
Spasticity is an umbrella term for impairments of muscle tone and control in people with damage to the brain and spinal cord. It is highly prevalent and results in pain, stiffness, and contribute to difficulties in activities of daily living. Current treatment options are limited, and many people experience only partial reduction in spasticity and frequent repeated treatments are needed.

Cryoneurolysis is a medical technique which involves the controlled freezing of the nerves. It has been approved in the UK for the treatment of pain in the context of spasticity through the targeting of nerves which control problematic muscles. Oxford University Hospitals NHS Foundation Trust has been offering this treatment routinely since January 2024. This pilot study aims to improve the understanding of the potential effectiveness of this treatment and its potential side effects when compared with a more commonly used treatment (Botulinum Toxin).

Participants will be randomly allocated to receive usual care with Botulinum Toxin (control group) or usual care with Cryoneurolysis (intervention group). The investigators will assess pain, goal attainment, side effects, spasticity, disability and independence in daily activities, and movement of the arm and leg. Assessments will be at baseline and then 6-, 12-, 18-, and 24-weeks following treatment. Participants who are randomised to the control group will have the opportunity to receive cryoneurolysis treatment after the 12 week follow up assessment.

The results of this study will help to guide future studies to examine the effectiveness of this treatment.

DETAILED DESCRIPTION:
Spasticity is an umbrella term for impairments of muscle activity and control in the context of damage or dysfunction in the central nervous system, occurring in up to 87% of spinal cord injury patients, 42% of stroke patients, and 80% of patients with multiple sclerosis. Spasticity results in pain, stiffness, and restrictions to activity including difficulties in personal care and mobility and a significant impact on quality of life.

Treatments including oral medications, botulinum toxin injections, and physical therapies can provide some degree of relief, but effectiveness varies widely. Many patients experience only partial reduction in spasticity, contributing to ongoing functional limitations. Botulinum toxin injections provide temporary relief necessitating frequent treatments (every 3-4 months). This is burdensome for patients and healthcare providers, with associated time and treatment costs. Pharmacological treatments can lead to systemic side effects including drowsiness, dizziness, and cognitive impairments. Surgical interventions are resource-intensive and require specialised medical facilities. Their associated costs, in terms of financial resources and healthcare infrastructure, significantly limit access for certain patients.

Cryoneurolysis, a novel medical technique, involves the controlled freezing of nerve tissue to temporarily disrupt its function. While primarily used for pain, there is a growing interest in its application for managing spasticity and it is currently approved for the treatment of pain in the context of spasticity at Oxford University Hospitals NHS Trust. Observational studies suggest immediate relaxation of the affected muscles, resulting in improved joint range of motion, enhanced functional mobility, and reduced pain. The investigators' own open-label proof-of-principle clinical data suggest the potential for substantial improvements in the impact of spasticity on quality of life.

This pilot randomised controlled study aims to improve the understanding of the potential clinical effectiveness and side effect profile of cryoneurolysis as a treatment for pain in the context of spasticity in people with a range of neurological conditions (e.g. acquired brain injury (ABI), spinal cord injury, stroke, multiple sclerosis).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial OR a positive opinion from a consultee is provided by a family member or carer (relative or friend) willing to provide personal consultee (PC) advice.
* Male or Female, aged 18 years or above.
* Diagnosed with a central neurological condition, including acquired brain injury (e.g. from ischaemic stroke, trauma, or haemorrhage), multiple sclerosis, and spinal cord injury.
* Clinical indication for Botulinum Toxin and Cryoneurolysis treatment, including pain associated with spasticity and with a clinically meaningful response to diagnostic nerve block to specific nerves or nerve branches that can be treated with cryoneurolysis.
* At least one rehabilitation goal related to management of pain resulting from spasticity.

Exclusion Criteria:

* Participant has received Botulinum toxin or cryoneurolysis within the last 90 days.
* Raynaud's syndrome.
* Cryoglobulinaemia.
* Cold urticaria.
* Bleeding disorders.
* Localised infection at intended treatment site.
* Planned oral antispasmodic medication dose changes.
* Pregnancy, breastfeeding, or planning pregnancy in the trial period.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who are currently enrolled in another trial may be excluded if it is deemed (in the investigator's opinion) that participation could influence the results for either study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scale | 6-weeks post-treatment
  An individualised outcome measure involving goal selection and goal scaling that is standardised in order to calculate the extent to which a patient's goals are met. GAS comprises of goals divided into a 5-point scale of level of expected outcome: from -2 (much less than expected) to +2 (much more than expected).

SECONDARY OUTCOMES:
Self-reported Pain | 6, 12, 18, and 24 weeks post-treatment
  Self-report, as measured by a numerical rating scale (range 0 - 10, higher scores indicating higher pain levels).
Douleur Neuropathique en 4 (DN4) | 6, 12, 18, and 24 weeks post-treatment
  Questionnaire used to determine whether pain is neuropathic in origin (range 0 - 10; a score of 4 or more suggests the presence of neuropathic pain).
Neuropathic Pain Symptom Inventory (NPSI) | 6, 12, 18, and 24 weeks post-treatment
  Questionnaire used to quantify neuropathic pain (range 0 - 100, higher scores reflect worse neuropathic pain).
Side Effects | 6, 12, 18, and 24 weeks post-treatment
  As measured by self-report side effects questionnaire
Goal Attainment Scale | 12-weeks post treatment
  An individualised outcome measure involving goal selection and goal scaling that is standardised in order to calculate the extent to which a patient's goals are met. GAS comprises of goals divided into a 5-point scale of level of expected outcome: from -2 (much less than expected) to +2 (much more than expected).
Modified Ashworth Scale | 6- and 12-weeks post treatment
  Assessment which requires the researcher to passively move the person's affected limb(s) and assess their resistance to movement (score range 0 - 4, higher score indicating increased in tone).
Modified Tardieu Scale | 6- and 12-weeks post treatment
  Assessment which requires the researcher to passively move the person's affected limb(s) and assess their resistance to movement (score range 0 - 4, higher score indicating increased resistance).
Spasticity | 6- and 12-weeks post treatment
  Directly assessed by measuring the muscle activity to a passive stretch
Range of Motion | 6- and 12-weeks post treatment
  Assessed using a goniometer
Patient Reported Impact of Spasticity Measure (PRISM) | 6- and 12-weeks post treatment
  Questionnaire assessing spasticity related quality of life (41 items that describe impacts of spasticity, each of which is rated on a scale of 0-4 from "never true for me" to "very often true for me").
EQ5D | 6- and 12-weeks post treatment
  Questionnaire assessing quality of life across 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels which are scored 1 - 5, with higher scores indicating worse outcome.
Spasticity Related Quality of Life instrument (SQoL-6D) | 6- and 12-weeks post treatment
  Questionnaire assessing spasticity related quality of life (range 0 - 24, higher score indicating worse condition)
Barthel Index | 6- and 12-weeks post treatment
  Scale measuring a person's ability to complete activities of daily living (range 0 - 100, higher scores indicating more independence)
Gait assessment - Walking Speed | 6- and 12-weeks post treatment
  Kinematic assessment of lower extremity function, using EMG and motion capture cameras. Walking speed is measured in meters per second (m/s), with slower speed indicating worse outcome.
Gait assessment - Gait profile score | 6- and 12-weeks post treatment
  Kinematic assessment of lower extremity function using EMG and motion capture cameras. The gait profile score is measured in degrees, with higher scores indicating more abnormality, and no maximum score.
Leg Activity Measure (LEG-A) | 6- and 12-weeks post treatment
  Questionnaire assessing lower extremity function (3 sections: Section A range: 0-36; Section B range 0-60; Section C range 0 - 36. Higher score indicates more difficulty/severity.)
Shriners Hospital Upper Extremity Evaluation (SHUEE) | 6- and 12-weeks post treatment
  Kinematic assessment of upper extremity function using motion capture cameras.
Arm Activity Measure (ARM-A) | 6- and 12-weeks post treatment
  Questionnaire assessing upper extremity function (2 sections: Section A range: 0-32; Section B range 0-52. Higher score indicates more difficulty.)
Functional Assessment Test for Upper Limb (FAST-UL) | 6- and 12-weeks post treatment
  Assessment of upper extremity function (selected movements assessed and scored between 0 - 3, with higher scores indicating ability to complete movement more fully).
Pressure Pain Thresholds (PPT) | 6, 12, 18, and 24 weeks post-treatment
  Sensory testing using a manual algometer to assess pain thresholds.

OTHER OUTCOMES:
Feedback Questionnaire/Interview | 24 weeks post treatment
  Qualitative feedback using either a semi-structured interview or a self-reported questionnaire (using the same questions as interview schedule), as per preference of participant, used to explore the satisfaction, experience, and anticipated barriers/facilitators to clinical implementation for the treatments.
Sleep Condition Indicator | 6, 12, 18, and 24 weeks post-treatment
  Questionnaire assessing self-reported insomnia symptoms (range 0-32, higher numbers indicate less symptoms of insomnia)
Goal Attainment Scale | 18- and 24-weeks post-treatment
  An individualised outcome measure involving goal selection and goal scaling that is standardised in order to calculate the extent to which a patient's goals are met. GAS comprises of goals divided into a 5-point scale of level of expected outcome: from -2 (much less than expected) to +2 (much more than expected).
Modified Ashworth Scale | 18- and 24-weeks post-treatment
  Assessment which requires the researcher to passively move the person's affected limb(s) and assess their resistance to movement (score range 0 - 4, higher score indicating increased in tone).
Modified Tardieu Scale | 18- and 24-weeks post-treatment
  Assessment which requires the researcher to passively move the person's affected limb(s) and assess their resistance to movement (score range 0 - 4, higher score indicating increased resistance).
Spasticity | 18- and 24-weeks post-treatment
  Directly assessed by measuring the muscle activity to a passive stretch
Range of motion | 18- and 24-weeks post-treatment
  Assessed using a goniometer
Patient Reported Impact of Spasticity Measure (PRISM) | 18- and 24-weeks post-treatment
  Questionnaire assessing spasticity related quality of life (41 items that describe impacts of spasticity, each of which is rated on a scale of 0-4 from "never true for me" to "very often true for me")
EQ5D | 18- and 24-weeks post-treatment
  Questionnaire assessing quality of life across 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels which are scored 1 - 5, with higher scores indicating worse outcome.
Spasticity Related Quality of Life instrument (SQoL-6D) | 18- and 24-weeks post-treatment
  Questionnaire assessing spasticity related quality of life (range 0 - 24, higher score indicating worse condition)
Barthel Index | 18- and 24-weeks post-treatment
  Scale measuring a person's ability to complete activities of daily living (range 0 - 100, higher scores indicating more independence)
Leg Activity Measure (LEG-A) | 18- and 24-weeks post-treatment
  Questionnaire assessing lower extremity function (3 sections: Section A range: 0-36; Section B range 0-60; Section C range 0 - 36. Higher score indicates more difficulty/severity.)
Arm Activity Measure (ARM-A) | 18- and 24-weeks post-treatment
  Questionnaire assessing upper extremity function (2 sections: Section A range: 0-32; Section B range 0-52. Higher score indicates more difficulty.)

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Centre for Enablement (OUH NHS-FT), Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified data are available upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Following publication of results
Access Criteria: Available upon reasonable request

REFERENCES:
- [Background] Wissel J, Manack A, Brainin M. Toward an epidemiology of poststroke spasticity. Neurology. 2013 Jan 15;80(3 Suppl 2):S13-9. doi: 10.1212/WNL.0b013e3182762448. PMID 23319481
- [Background] Winston P, Mills PB, Reebye R, Vincent D. Cryoneurotomy as a Percutaneous Mini-invasive Therapy for the Treatment of the Spastic Limb: Case Presentation, Review of the Literature, and Proposed Approach for Use. Arch Rehabil Res Clin Transl. 2019 Oct 17;1(3-4):100030. doi: 10.1016/j.arrct.2019.100030. eCollection 2019 Dec. PMID 33543059
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Turner-Stokes L, Jacinto J, Fheodoroff K, Brashear A, Maisonobe P, Lysandropoulos A, Ashford S; Upper Limb International Spasticity (ULIS-III) study group. Longitudinal goal attainment with integrated upper limb spasticity management including repeat injections of botulinum toxin A: Findings from the prospective, observational Upper Limb International Spasticity (ULIS-III) cohort study. J Rehabil Med. 2021 Feb 24;53(2):jrm00157. doi: 10.2340/16501977-2801. PMID 33616192
- [Background] Skoog B, Jakobsson KE. Prevalence of Spasticity and Below-Level Neuropathic Pain Related to Spinal Cord Injury Level and Damage to the Lower Spinal Segments. J Rehabil Med Clin Commun. 2020 Mar 8;3:1000039. doi: 10.2340/20030711-1000039. eCollection 2020. PMID 33884141
- [Background] Rizzo MA, Hadjimichael OC, Preiningerova J, Vollmer TL. Prevalence and treatment of spasticity reported by multiple sclerosis patients. Mult Scler. 2004 Oct;10(5):589-95. doi: 10.1191/1352458504ms1085oa. PMID 15471378
- [Background] Kim PS, Ferrante FM. Cryoanalgesia: a novel treatment for hip adductor spasticity and obturator neuralgia. Anesthesiology. 1998 Aug;89(2):534-6. doi: 10.1097/00000542-199808000-00036. No abstract available. PMID 9710418
- [Background] Biel E, Aroke EN, Maye J, Zhang SJ. The applications of cryoneurolysis for acute and chronic pain management. Pain Pract. 2023 Feb;23(2):204-215. doi: 10.1111/papr.13182. Epub 2022 Dec 4. PMID 36370129
- [Background] Bhimani R, Anderson L. Clinical understanding of spasticity: implications for practice. Rehabil Res Pract. 2014;2014:279175. doi: 10.1155/2014/279175. Epub 2014 Sep 4. PMID 25276432